CLINICAL TRIAL: NCT02668718
Title: Adjuvant Radiation Therapy vs. Watchful Waiting in Prostate Cancer Patients With Positive Margins or Capsular Penetration After Radical Prostatectomy
Brief Title: Adjuvant Radiation Therapy vs. Watchful Waiting Following Radical Prostatectomy in High Risk Prostate Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Teuvo Tammela, M.D., Ph.D., Professor of Surgery, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FP-FINROG-0301
Record Dates: First submitted 2016-01-27; First posted 2016-01-29 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Prostatic Neoplasms
Keywords: radiotherapy, adjuvant; prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adjuvant radiotherapy (Other): Patients who were randomized to adjuvant radiotherapy following radical prostatectomy
  Interventions: Radiation: Adjuvant radiotherapy
- Watchful waiting (No Intervention): Patients who were randomized to watchful waiting following radical prostatectomy

INTERVENTIONS:
Radiation: Adjuvant radiotherapy — The radiation therapy will be given in 37 fractions of 1.8 Gy per day, five days per week. The total dose of radiation will be 66.6 Gy.
  Arms: Adjuvant radiotherapy

SUMMARY:
The purpose of this study is to determine whether adjuvant radiotherapy following radical prostatectomy in prostate cancer patients with positive margins or capsular penetration improves biochemical, overall and/or cancer specific survival and whether adjuvant radiotherapy is reasonably well tolerated when compared to watchful waiting.

DETAILED DESCRIPTION:
In this study the investigators will evaluate adjuvant radiation therapy vs. watchful waiting in prostate cancer patients with positive margins or capsular penetration after radical prostatectomy. This is a randomized, open label, multicentre, collaborative study of FinnProstate Group and Finnish Radiation Oncology group.

ELIGIBILITY:
Inclusion Criteria:

Patients with pT3aN0M0 or pT2N0M0 prostate cancer with a positive margin, gleason score 2-10, preoperative PSA < 20 ug/l, postoperative PSA <0.5 ug/l after surgery (within 8 weeks), the WHO performance status 0-2, life expectancy at least 3 months, informed consent obtained.

Exclusion Criteria:

Other simultaneous cancer therapy including systemic endocrine therapy; more than 12 weeks has elapsed since surgery for prostate cancer; metastatic disease (N+ or M1); cancer invasion to the seminal vesicles; any other previous malignancy within the last 5 years except basalioma or squamous cell carcinoma of the skin; any contraindication to irradiation (severe locoregional infection, prior radiation therapy to the prostate/bladder); any physical or mental condition, which in the opinion of the investigator, may interfere with patient's ability to comply with scheduled visits.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2004-03; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Biochemical disease-free survival | Five years
Overall survival | Five years
Cancer specific survival | 5 years

SECONDARY OUTCOMES:
Local recurrence verified by needle or surgical biopsy | Five years
Adverse events | Five years

CONTACTS AND LOCATIONS:
Overall Officials: Teuvo Tammela, M.D., Ph.D., Principal Investigator — Tampere University Hospital

IPD SHARING:
Plan to Share IPD: Undecided